CLINICAL TRIAL: NCT00271492
Title: Endothelin in the Coronary Circulation in Early Atherosclerosis in Humans
Brief Title: Correlation of Endothelial Function and Early Coronary Artery Disease in Humans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Amir Lerman, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 48-99
Record Dates: First submitted 2005-12-29; First posted 2006-01-02 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Endothelial Dysfunction
MeSH Terms: interventions — Atrasentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Active Comparator): Qualifying patients took Atrasentan, 1 pill per day for 6 months, to determine if it had a favorable affect on patients who took it over those who were randomized to placebo.
  Interventions: Drug: Atrasentan
- 2 (Placebo Comparator): placebo group to be compared to the actual medication
  Interventions: Drug: atrasentan

INTERVENTIONS:
Drug: Atrasentan — 1 10mg capsule to be taken daily for 6 month study period.
  Other Names: Xinlay
  Arms: I
Drug: Atrasentan — 1 10mg capsule per day for the 6 month study period.
  Other Names: Xinlay
  Arms: I
Drug: atrasentan — One 10 mg capsule per day for 6 month study period
  Other Names: Xinlay
  Arms: 2

SUMMARY:
Qualifying patients who are scheduled for angiogram with endothelial function testing are approached to participate in this protocol (consent form reviewed with patient). Those who are willing to participate will have additional measurements taken during their angiogram as part of this protocol. Patients who are diagnosed with Endothelial Dysfunction as a result of a clinically indicated angiogram will be eligible to participate in a 6 month medication trial (Atrasentan vs. placebo - randomized, blinded trial). Patients are monitored closely during the 6 month trial via phone calls and blood testing for assessment. At the end of the 6 months they return to Mayo for a repeat angiogram to assess endothelial function for any changes or improvements.

DETAILED DESCRIPTION:
Aim I: To determine the activity of the endogenous endothelin system in the coronary circulation in humans with coronary endothelial dysfunction and atherosclerosis risk factors. Aim II: To assess the potential of chronic endothelin receptor antagonists to improve preexisting coronary endothelial dysfunction and myocardial perfusion in humans and Aim III: To assess the effect of chronic endothelin receptor antagonism on the endogenous nitric oxide system in association with oxidative stress in humans with early coronary disease risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 85 years
* Male or female

Exclusion criteria:

* Left dominant circulation
* Heart failure with EF <40%
* Unstable angina
* MI or angioplasty of the LAD or circumflex with 6 months prior to entry into the study
* Use of radiographic contrast agent within 12 hours of entry into the study
* Use of investigational agents within one month of entry into the study
* Patients who require treatment with positive inotropic agents other than digoxin during the study
* Patients with cerebrovascular accident within 6 months prior to entry into the study
* Significant endocrine, hepatic, renal disorders; local or systemic infectious disease within 4 weeks prior to entry into study
* Pregnancy or lactation
* Mental instability
* Federal Medical Center patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2001-07; Primary Completion 2006-06 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To find out what effects (good and bad) the medication Atrasentan has on the heart | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Reriani M, Raichlin E, Prasad A, Mathew V, Pumper GM, Nelson RE, Lennon R, Rihal C, Lerman LO, Lerman A. Long-term administration of endothelin receptor antagonist improves coronary endothelial function in patients with early atherosclerosis. Circulation. 2010 Sep 7;122(10):958-66. doi: 10.1161/CIRCULATIONAHA.110.967406. Epub 2010 Aug 23. PMID 20733096